CLINICAL TRIAL: NCT03966001
Title: Formation of the Cesarean Scar Defect After the First Cesarean. A Prospective Observational Study of Planned Versus Emergency Cesarean Sections
Brief Title: Cesarean Scar Defect Formation After First Cesarean Section.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Adnan Orhan, Medical Doctor, Researcher, Obstetrician and Gynecologist, Uludag University
Other Study IDs: UU-SUAM-2019-8/34
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Cesarean Section Complications; Cesarean Wound Disruption; Cesarean Wound; Dehiscence
Keywords: Cesarean scar pregnancy; Isthmocele; Uterine niche; Cesarean scar defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Planned Cesarean Group: Pregnant women undergoing a planned cesarean section at 38-42 gestational week.
  Interventions: Other: Transvaginal sonography at six months after cesarean section; Other: Transvaginal sonography at twelve months after cesarean section
- Emergency Cesarean Group: Pregnant women who are planning to give normal birth between 38-42 weeks of gestation but have to been performed an urgent cesarean section due to an emergency such as acute fetal distress, cephalo-pelvic disproportion or another obstetrical condition.
  Interventions: Other: Transvaginal sonography at six months after cesarean section; Other: Transvaginal sonography at twelve months after cesarean section

INTERVENTIONS:
Other: Transvaginal sonography at six months after cesarean section — In the sixth month after cesarean section, Women in both groups will undergo a detailed pelvic examination and transvaginal ultrasonographic evaluation for the cesarean scar defect.
  Other Names: Transvaginal sonography 6th month after C/S
Other: Transvaginal sonography at twelve months after cesarean section — In the twelfth month after cesarean section, Women in both groups will undergo a detailed pelvic examination and transvaginal ultrasonographic evaluation for the cesarean scar defect.
  Other Names: Transvaginal sonography 12th month after C/S

SUMMARY:
This study is a prospective observational study which will monitor how cesarean section in the first pregnancy will develop a cesarean scar defect. Patients with planned cesarean section in their first pregnancy and those with an emergency cesarean section will be monitored for one year.

DETAILED DESCRIPTION:
Cesarean scar defects, which may develop after cesarean deliveries, are associated with menstrual bleeding problems, infertility, and poor obstetric outcomes. No matter how excellent and standard surgical technique is applied, scar defects may develop after cesarean section. However, when cesarean operation decision is taken, the existing operational conditions can affect the formation of cesarean scar defect in the future. Although the surgical technique is the same, a planned cesarean operation and an emergency cesarean section may differ for a future cesarean scar defect that may develop in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18-45-year-old patients
* Patients who have undergone a planned or emergency cesarean section within the 38-42th gestational week.

Exclusion Criteria:

* Spontaneous vaginal birth
* Preterm birth
* Pregnant women with an obstetrical or gynecological complication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women at 38-42th gestational weeks.
Study Population: The study population consists of pregnant patients who are in their 38-42th gestational weeks and who undergo planned or emergency cesarean section.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Cesarean Scar Defect (Niche) | 10 minutes
  The presence of a "niche" at the site of cesarean delivery scar diagnosed at the time of transvaginal ultrasonography

SECONDARY OUTCOMES:
Postmenstrual spotting | 7-10 days
  Any vaginal bleeding that occurs after the usual menstrual period.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Director — Uludag University Hospital, 16059, Bursa, Turkey; Bilge Cetinkaya Demır, Assoc.Prof., Principal Investigator — Uludag University Hospital, 16059, Bursa, Turkey
Locations (1):
- Uludag University Hospital, Department of Obstetrics and Gynecology, Bursa, Ozluce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within nine months after the study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requesters will be required to sign a data access agreement form.
URL: http://www.uludag.edu.tr

REFERENCES:
- [Background] Antila-Langsjo R, Maenpaa JU, Huhtala H, Tomas E, Staff S. Comparison of transvaginal ultrasound and saline contrast sonohysterography in evaluation of cesarean scar defect: a prospective cohort study. Acta Obstet Gynecol Scand. 2018 Sep;97(9):1130-1136. doi: 10.1111/aogs.13367. Epub 2018 May 29. PMID 29754409
- [Background] Setubal A, Alves J, Osorio F, Guerra A, Fernandes R, Albornoz J, Sidiroupoulou Z. Treatment for Uterine Isthmocele, A Pouchlike Defect at the Site of a Cesarean Section Scar. J Minim Invasive Gynecol. 2018 Jan;25(1):38-46. doi: 10.1016/j.jmig.2017.09.022. Epub 2017 Oct 9. PMID 29024799
- [Background] Cali G, Timor-Tritsch IE, Palacios-Jaraquemada J, Monteaugudo A, Buca D, Forlani F, Familiari A, Scambia G, Acharya G, D'Antonio F. Outcome of Cesarean scar pregnancy managed expectantly: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Feb;51(2):169-175. doi: 10.1002/uog.17568. PMID 28661021
- [Result] Antila-Langsjo RM, Maenpaa JU, Huhtala HS, Tomas EI, Staff SM. Cesarean scar defect: a prospective study on risk factors. Am J Obstet Gynecol. 2018 Nov;219(5):458.e1-458.e8. doi: 10.1016/j.ajog.2018.09.004. Epub 2018 Sep 18. PMID 30240650
- [Result] Ades A, Parghi S. Laparoscopic Resection of Cesarean Scar Ectopic Pregnancy. J Minim Invasive Gynecol. 2017 May-Jun;24(4):533-535. doi: 10.1016/j.jmig.2016.11.006. Epub 2016 Nov 17. PMID 27867050